CLINICAL TRIAL: NCT02976974
Title: Efficacy of Manual Therapy and Therapeutic Exercise in Patients With Shoulder Adhesive Capsulitis. Which Factors Are More Correlated With?
Brief Title: Efficacy of Manual Therapy and Exercise in Patients With Shoulder Adhesive Capsulitis. A Randomized Clinical Trial.
Acronym: MTEAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Malaga (Other)
Responsible Party: Principal Investigator, Alejandro Luque-Suarez, Efficacy of manual therapy and exercise in patients with shoulder adhesive capsulitis. Which biomechanics/psychological factors are more correlated with?, University of Malaga
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMA MTEAC
Record Dates: First submitted 2016-11-22; First posted 2016-11-30 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Shoulder Pain
Keywords: chronic pain; central sensitization; function; force; ultrasonography
MeSH Terms: conditions — Shoulder Pain; Chronic Pain | interventions — Musculoskeletal Manipulations; Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy (MT) (Experimental): MT: Manual Therapy. Application of different manual therapy techniques through posterior and inferior humeral head slides, as well as scapular movements. Also, rotator interval stretching will be done.
  Interventions: Other: Manual therapy
- Therapeutic exercise (E) (Experimental): E: Therapeutic Exercise.
  Shoulder extension: Elastic bands. Shoulder flexion: Elastic bands Shoulder external rotation: Elastic bands. Scapulothoracic stability: Movement of scapular adduction guided by the physiotherapist, keeping the position for few seconds ; standing "push up" on the wall.
  Thoracic column movements: Flexion-extension
  Interventions: Other: Manual therapy; Other: Therapeutic exercise

INTERVENTIONS:
Other: Manual therapy — Application of different manual therapy techniques through posterior and inferior humeral head slides, as well as scapular movements. Also, rotator interval stretching will be done.
Other: Therapeutic exercise — * Shoulder extension: Elastic bands.
  * Shoulder flexion: Elastic bands
  * Shoulder external rotation: Elastic bands.
  * Scapulothoracic stability: Movement of scapular adduction guided by the physiotherapist, keeping the position for few seconds ; standing "push up" on the wall.
  * Thoracic column movements: Flexion-extension
  Arms: Therapeutic exercise (E)

SUMMARY:
The efficacy of manual therapy and therapeutic exercise in patients suffering from adhesive capsulitis of the shoulder will be studied. Furthermore, different biomechanic and psychosocial factors will be measured with a nine month follow-up

DETAILED DESCRIPTION:
Adhesive capsulitis of the shoulder is a painful entity characterized by stiffness in the shoulder joint. There exist different clinical trial related to this pathology, however a lack of information of both efficacy and methodology used in manual therapy treatment remains unclear, as well as therapeutic exercise treatment. Furthermore, the duration of the improvement after different conservative treatments is also unknown. Besides, little is known about which factors are more correlated with pain and function.Thus, biomechanic and psychosocial factors together with ultrasound measurements and blood glucose concentration (see "outcome and secondary measures" section ) will be analyzed before and after the treatment, with a nine months follow up. Results will be spread showing short term effects and long term effects in different publications.

Hence, the aim of this study is twofold: i)To analyze the efficacy of manual therapy and therapeutic exercise in patients with shoulder adhesive capsulitis; ii) To correlate pain and function with ultrasonography, biomechanic and psychosocial factors, as well as blood glucose concentration, before and after the treatments proposed with a nine months follow up.

Method

This study is designed as a clinical trial, with two randomised parallel groups comparing two different conservative intervention (MT vs MT+E) (See "Arms and Interventions" section). It will be carried out in different Hospital and primary care centers where patients suffering from adhesive capsulitis of the shoulder will be asked to participate in the project. If participants are eligible then they will be include in the study. All participants will have to sign informed consent after be shown about the whole project as by written (informative sheet) as by speech from the physiotherapist in charge.

Once include in the study definitely, all factors detailed (see "outcome measures" section) will be measured. Also, every factor will be correlated with shoulder pain and function. This way, the investigators could predict which factor are more correlated with. Furthermore, if significant correlations are found, such factors could be used as predictors or monitoring tool when patients with shoulder adhesive capsulitis are treated

ELIGIBILITY:
Inclusion Criteria:

* People suffering from adhesive capsulitis as indicated by passive range of motion loss >25% in at least 2 movement planes, together with at least 50% loss of passive external rotation in comparison with the uninvolved shoulder.

Exclusion Criteria:

* Shoulder pain that was deemed to be originating from any passive and/or neck movement or if there was a neurological impairment, osteoporosis, haemophilia and/or malignancies
* Corticoid injections during the six months prior to the study
* Analgesic-antiinflammatory medication intake during the intervention phase of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-07-30 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline SPADI (Shoulder Pain And Disability Index) questionnaire at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  The Shoulder Pain and Disability Index (SPADI) is a self-administered questionnaire that consists of two dimensions, one for pain and the other for functional activities.

SECONDARY OUTCOMES:
Change from baseline pressure algometry at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Assessment of central sensitization:
  It will be carried out on the affected and unaffected shoulder (mid belly of medium deltoid muscle: 2 cm under acromion). Also, the quadriceps rectus femoris (ipsilateral to frozen shoulder, middle spine iliac antero-superior (SIAS) and top patella) will be assessed.
Change from baseline ultrasonography at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Different structures will be measured by ultrasonography such as tendons (supraspinatus, infraspinatus, subscapularis and long head biceps tendon) and ligaments (coracohumeral and upper glenohumeral ligaments). Furthermore, acromiohumeral distance and coracohumeral distance will be analyzed. In addition, presence of neovascularization will be studied.
Change from baseline electromyography at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  It will be investigated the surface electromyographic (EMG) relative muscle activity of the upper (UT) and lower trapezius (LT) as well as serratus anterior (SA) muscles during both ascending and descending phases of arm elevation in participants with adhesive capsulitis of the shoulder
Change from baseline dynamometry at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Assessment of shoulder force (unit of measure: kilograms) in seated position (handheld dynamometer) :
  * Elevation in the scapular plane at 90°
  * Outer rotation with flexion elbow at 90°
  * Inner rotation with flexion elbow at 90°
  * Lift off position: Patient places arm behind the back, 90° flexion elbow.
  Three measurements will be carried out in each position. The mean will be the final value.
Change from baseline blood glucose concentration at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  To assess metabolic factors venous blood samples will be collected.Information about a person's average levels of blood glucose, over the past 3 months (A1C) will be obtained with the "A1C" test or glycohemoglobin test.
Change from baseline range of movement (ROM) at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Measurement of mobility in different planes:
  Active shoulder flexion and abduction will be measured with the patient seated, in the scapular plane and relative to the thorax. In addition, active external and internal rotation will be measured in neutral (shoulder in adduction), 30°, 60° and 90° of abducted position.
Change from baseline heart rate variability (HRV) at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Measurement of Autonomic nervous system activity:
  Resting HRV provides quantitative information regarding cardiac autonomic tone.
Change from baseline CSI questionnaire at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Measurement of central sensitization (CS):
  The Central Sensitization Inventory (CSI) was developed to assess the overlapping health-related symptom dimensions of CS
Change from baseline "pain vigilance and awareness" questionnaire at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  The Pain Vigilance and Awareness Questionnaire(PVAQ) is a 16-item measure of pain-related awareness and vigilance. It shows predicted relations with measures of attention-related pain coping strategies, supporting the validity of the total score as a measure of attention to pain
Change from baseline pain Catastrophizing Scale questionnaire at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Assessment of the mechanisms by which catastrophizing impacts on pain experience.
Change from baseline short form-36 (SF-36) at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Measurement of Quality of life:
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.
Change from baseline McGill questionnaire at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Measurement of pain:
  The McGill Pain Questionnaire can be used to evaluate a person experiencing significant pain. It can be used to monitor the pain over time and to determine the effectiveness of any intervention.
Change from baseline Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Assessment of quality of life.:
  This questionnaire measure upper limb symptoms as well as patient ability to do certain activities.
Change from baseline Autonomic Symptom Profile questionnaire (ASP) at nine months | time (t) 1(prior to treatment), t2 (just received treatment), t3 (3 months later), t4 (6 months later), t5 (9 months later)
  Measurement of Autonomic nervous system activity:
  The Autonomic Symptom Profile (ASP) is a validated self-report questionnaire that comprehensively assesses autonomic symptoms across 11 subscales and yields a composite autonomic symptom score

CONTACTS AND LOCATIONS:
Overall Officials: ALEJANDRO LUQUE-SUAREZ, PT, PhD, Principal Investigator — UNIVERSITY OF MALAGA, SPAIN
Locations (3):
- Spain (3):
  - Las Albarizas primary care centre, Fuengirola, Malaga
  - Las Lagunas Care Centre, Fuengirola, Malaga
  - San Pedro primary care centre, Marbella, Malaga

IPD SHARING:
Plan to Share IPD: Yes
The results obtained in this project will be disseminated to the research community through different vias such as publications and oral/poster presentations